CLINICAL TRIAL: NCT02008552
Title: Research for Genetic Factors Involved in the Individual Susceptibility to Develop a Valvulopathy During a Medicinal Exposure in the Benfluorex.
Brief Title: Study of the Effect of the Benfluorex
Acronym: MEDIAGENE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MEDIAGENE
Record Dates: First submitted 2013-11-28; First posted 2013-12-11 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Blood Sample
Keywords: Genetic factor; Valvulopathy; Mediator
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mediagene (Other): Sampling blood
  Interventions: Genetic: Sampling of blood

INTERVENTIONS:
Genetic: Sampling of blood — Sampling of blood was taken and analyse to research factor genetic

SUMMARY:
More than 5 million persons in France exposed, in last years, to the taking of the Benfluorex.

Arisen, at certain patients, of a valvulopathy characterized by mitrals and/or aortic leaks Withdrawal of the French market: nov. 2009 Only a percentage limited by exposed patients developed a severe valvulopathy (1/1000), whereas on the contrary, many patients were exposed during years without developing the slightest anomaly.

The hypothesis is the existence of a particular genetic susceptibility at the patients having developed a valvulopathy continuation in the exposure in this medicine.

Existence of one varying genetics with strong effect. The purpose is to identify involved genetic factors.

ELIGIBILITY:
Inclusion Criteria of the cases :

* Individual presenting a typical medicinal valvulopathy defined by:
* A previous exposure of at least 6 months in the benfluorex or occasional exposure accepted about is the posology. The preliminary exposure in the dexfenfluramine or in the fenfluramine is authorized.
* A picture board of insufficiency mitral restrictive and/or aortic restrictive (in echocardiography) typical of a medicinal achievement, a gravity (rank I - IV), without cause associated of valvulopathy with compatible macroscopic and histological aspect (for the operated patients).
* Individual followed in one of the sites of study or recruited via associations AVIM and CADUS.
* Individual of Caucasian origin
* Individual having signed the form of specific consent for the study individual .

Inclusion criteria of witnesses :

* Individual presenting an exposure previous to the benfluorex superior or equal to the equivalent of 2 years of treatment in 3 tablets a day and pursued to 2 years preceding the realization of a cardiac echography of screening. The preliminary exposure in the dexfenfluramine or in the fenfluramine is authorized.
* Individual presenting a strictly normal cardiac echography in particular: absence of valvulopathy significant, of morphological valvular anomaly (event without echography) and of valvular, including "trivial" leak at the aortic level. The mitrals micro leaks "physiological" are accepted.
* Individual having been seen for screening in one of the sites of study or in in French firms cardilogie which cardiologists are members of the French Society of Cardiologyor or via the law firms of the civil parties or having been included in the forward-looking study coordinated by Pr. TRIBOUILLOY (which the objective is to compare the echography data of a group of patients having been treated at least 3 months in the benfluorex and with a group of patients diabetics having never received this medicine).
* Individual of Caucasian origin.
* Individual having signed the form of specific consent for the study

Exclusion criteria of the cases:

* Individual presenting another associated heart disorder.
* Individual having been exposed to another agonists of the receivers 5-HT2B such as the pergolide, the cabergoline, the lisuride, the quibbled by-products or the ecstasy.
* Individual having explicitly refused to participate in the study.

Exclusion criteria of witnesses :

- Individual having explicitly refused to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2013-10-18 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
Identify the genetic factors | 12 months
  Identify the genetic factors involved in the individual susceptibility to develop a valvulopathy during a medicinal exposure in the benfluorex.

SECONDARY OUTCOMES:
Compare the quality of life | 12 months
  Compare the quality of life of the cases and the witnesses via the completion of Two validated questionnaires of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Irène Frachon, PH, Principal Investigator — CHRU de Brest
Locations (7):
- France (7):
  - Hôpital Sud Amiens, Amiens
  - CHRU de Brest, Brest
  - CHU de la Côte de Nacre Caen, Caen
  - Hôpital Saint Philibert, Lomme
  - Hôpital La Timone Marseille, Marseille
  - Institut du Thorax Nantes, Nantes
  - Faculté de médecine Toulouse, Toulouse